CLINICAL TRIAL: NCT05744284
Title: It is Time to Change Method of Skin Incision From Scalpel to Electrocautery.
Brief Title: Electrocautery for Safe Skin Incision
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Isidoro Di Carlo, MD, PhD, FACS, Professor, University of Catania
Other Study IDs: IDC-001
Record Dates: First submitted 2023-01-28; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Skin Injury
Keywords: Electrocautery; scalpel
MeSH Terms: interventions — Electrocoagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Sex, age, kind of disease in relation to the organ affected: Sex, age, kind of disease in relation to the organ affected and type of surgical procedure and related incision have been investigated. Patients with diabetes mellitus, coagulation disorders and those submitted to a treatment of steroids and anticoagulant; patients previously operated with scar in the site of the second operations, or with anemia or with active source of infection in any part of the body where excluded from the study.
  Interventions: Device: electrocautery

INTERVENTIONS:
Device: electrocautery — advantages reported in this study in terms of wound infections, healing time, postoperative pain and cosmetic results in association with economic gain for saving in the purchase of scalpels, represent a formidable motivation for the surgeons to abandon the scalpel in favors of diathermy

SUMMARY:
The use of electrocautery to incise the skin is still debated. Aim of the present study is to contribute at the use of electrocautery for skin incision as safe procedure both for patients and surgeons.

DETAILED DESCRIPTION:
All patients observed between 2016 and 2021 at the Department of Surgical Sciences, Organ Transplantation, and Advanced Technologies of University of Catania and submitted to abdominal surgery in which the incision of the skin have been done by electrocautery, have been considered. Sex, age, kind of disease in relation to the organ affected and type of surgical procedure and related incision have been investigated. Patients with diabetes mellitus, coagulation disorders and those submitted to a treatment of steroids and anticoagulant; patients previously operated with scar in the site of the second operations, or with anemia or with active source of infection in any part of the body where excluded from the study.

The ethical approval isn't necessary because is a retrospective study. All patients have express the oral informed consent to participate at this study.

In this retrospective study was analyzed the skin incision that has been classified into laparotomic or laparoscopic, in elective or emergency surgery. The laparotomic included large (large midline as xipho-umbilical or umbilical pubic incision, subcostals or pararectal) and small (small midline no more than 7 cm, inguinal, McBurney) skin incisions. The laparoscopic on the opposite involve incisions from minimum of 1 cm or less for introduction of trocars, and a maximum of 10 cm to extract organ. The subcutaneous layer has been closed using an interrupted suture using Vycril®3-0 on the opposite the skin suture has been done using metallic clips.

All patients have been submitted to general or spinal anesthesia. Antibiotic prophylaxis was done, following the guidelines related to the disease (5). Patients submitted to hernioplasty of laparoscopic cholecystectomy or any procedure in which the literature have reached a consensus any antibiotic treatment including the prophylaxis have not been done (5).

The outcomes considered are wound infections, post-operative pain, healing time, cosmetic results. The post operative pain has been related to the administration of paracetamole 1 gr every 12 hours for the first 3 days. The healing time and cosmetic results have been evaluated both during the hospitalization or in the out patients clinics, after 10 from surgical procedure at moment of ablation of metallic clips, and/or 20 days after the surgical incision with final clinical evaluations of the scar. Finally considering the medical records and operative reports, patients were contacted 6 months later by phone by resident in surgery ask them to evaluate their scar. The patient was asks simple to define their scar as acceptable and consequently patient satisfied or not acceptable so patient not satisfied.

We, also, consider the reported injury to surgeons or theater workers during the surgical procedure. Particularly we have reported the burns from hole in the gloves related to an absent respect of the isolated generator circuit

All patients were treat an expert surgeon, that used the same technique for the incision skin.

The skin incision has been done using the following rules: the cutting diathermy have been used to incise the skin. If bleeding comes from the dermis, the coagulation diathermy has been shortly used using the tip of the headpiece, without forceps. To incise the skin we have used a Valleylab force TX Medtronic Italy equipped with standard diathermy pen electrode, set on cutting mode for skin at 20 KHz sinusoidal current and on coagulation mode at K40 Hz both for skin and for deeper tissues (6).

Electrosurgery works by electrons' handling on living tissue using an alternating current density sufficient to create heat within tissue cells to destroy them.

It is mandatory to consider the mode of use electrosurgery. In the cutting mode, a continuous current produce extreme heat causing vaporization so the conversion of the cells into steam. When we use the electrosurgery unit into cutting mode for the skin the cells vaporize and the tissue is divided with a minimum devitalization, the thermal damage is minimal and it is not propagated to neighboring cells. Differently the coagulation mode that cause high thermal damage and necrosis of adjacent cells.

ELIGIBILITY:
Inclusion Criteria:

* surgical procedure with electrocautery skin incision

Exclusion Criteria:

* previews scars
* infections
* anemia

Max Age: 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: A total of 281 patients (119 females, 162 males) with a median age of 60 years were scheduled for abdominal surgery.
  Most of the patients have submitted to surgical procedures involving the small and large intestine (160 patients, 56.9%). Others patients were operated for liver, gallbladder, spleen or pancreas (41 patients, 14.5%), esophagus stomach or duodenum (4 patients, 1.4%) disease. Finally, some patients undergone to hernioplasty (57 patients, 20.2%). And at the least we have grouped as miscellaneous some patients undergoing procedures that concerned the subcutaneous or unspecified (19 patients, 6.7%).
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Wound infections | 10 days
  The wound infections were recorded in patients undergoing emergency surgery with laparotomic incisions. As sign of infection were observed fever, pain, hyperaemia and presence of pus.
Post-operative pain | 24 hours after procedures
  Patients refer pain classified as 1-2 in a numerical rating scale from 0 to 10, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
Cosmetic results | 6 months after surgery
  The patient was asked simple to define their scar as acceptable and consequently patient satisfied or not acceptable so patient not satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Isidoro Di carlo, Catania, CT, Italy

DOCUMENTS (1):
  • Study Protocol (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT05744284/Prot_000.pdf